CLINICAL TRIAL: NCT00713141
Title: Evaluation of Brain Function Before and After Standard Chemotherapy for Early Breast Cancer
Status: Completed | Type: Observational
Sponsor: National University Hospital, Singapore (Other)
Other Study IDs: BR03/09/04
Record Dates: First submitted 2008-07-10; First posted 2008-07-11 (Estimated); Last update posted 2010-08-31 (Estimated); Status verified 2010-08

CONDITIONS: Early Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional

GROUPS / COHORTS (1):
- 1: Early breast cancer

SUMMARY:
Primary Objective

* To investigate and clearly document the presence and extent of cognitive decline, if any, in women of Asian origin following standard-dose systematic adjuvant chemotherapy for the treatment of breast cancer
* Investigation and establishment of a relationship between degree of oxidative DNA and lipid damage as indicated by plasma and urinary biochemical markers.

Secondary Objective

• To validate the use of hydrogen peroxide and serum amyloid as biomarkers of damage

DETAILED DESCRIPTION:
As the survival rate and prognosis of cancer improve, there is increasing recognition of the presence of a long term negative impact of standard chemotherapy on cognition, namely in the domains of attention, memory, psychomotor speed and executive functions. The purported incidence varies between 10-50%, the mechanism is unknown and it is unclear who is at risk. This impact has also not been studied and documented in the Asian population.

This proposal outlines a study that intends to prospectively (1) investigate and document the incidence and severity of cognitive impairment following systemic chemotherapy for breast cancer in Asian women in the acute and prolonged setting, and (2) to relate these cognitive changes to damage to DNA and lipids (two major targets of attack by toxic agents) as indicated through tests conducted on blood and urine samples.

Thirty breast cancer patients who will be required to undergo standard chemotherapy will be recruited for a pilot study to determine the acceptability of the procedure and to establish the size of the effects under investigation. A 45-minute neurocognitive assessment will be administered at three time points: before commencement of chemotherapy, and at 6 months and 1 year following completion of chemotherapy. Blood and urine samples will be collected just prior to the commencement of chemotherapy, after the first cycle of chemotherapy, and also at 6 months and 1 year post completion of chemotherapy.

It is hypothesized that (1) there will be decrements in performance on the neurocognitive measures post-chemotherapy; (2) the presence of cognitive decline will correlate with the presence of markers of oxidative damage in the blood and urine samples. The benefits of this project are two fold. Firstly, it will allow research into and documentation of the possible presence of cognitive decline following chemotherapy in Asian women, which is important in allowing patients to make fully-informed consent with regard to treatment. Secondly, if a relationship between the presence of cognitive decline and the presence of biochemical markers of oxidative damage can be established, this can potentially lead to new treatment methods that may reduce the cognitive decline that has been associated with the chemotherapeutic process.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically documented breast cancer
2. Females greater than 18 years old
3. Eastern Cooperative Oncology Group (ECOG) Performance status 0,1,2
4. Requires to undergo standard-dose systemic adjuvant chemotherapy
5. Patients must be informed of nature of study and sign an informed consent form

Exclusion criteria

a. Dementia/significantly altered mental status that will prohibit the understanding and/or giving of informed consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A pilot study involving 30 women who have been diagnosed with breast cancer and will undergo standard adjuvant chemotherapy will be conducted first. This is to allow (1) the establishment of the acceptability of the procedure to patients and (2) documentation of the various effect sizes associated with (a) cognitive changes (b) changes in the level of the various biochemical markers following chemotherapy (c) the relationship between extent of cognitive decline and extent of DNA damage. It is estimated that up to approximately 100 patients can be recruited to participate in the main study.
Sampling Method: Probability Sample
Enrollment: 30
Dates: Start 2004-11

CONTACTS AND LOCATIONS:
Overall Officials: Chiung Ing Wong, MRCP, MB ChB, Principal Investigator — National University Hospital, Singapore
Locations (1):
- National University Hospital, Singapore, Singapore